CLINICAL TRIAL: NCT05524922
Title: A Registered Observational Cohort Study on Neurodegenerative Associated With Sleep Disorder.
Brief Title: A Registered Cohort Study on Neurodegenerative Associated With Sleep Disorder.
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort-Sleep Disorder
Record Dates: First submitted 2022-08-28; First posted 2022-09-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-09

CONDITIONS: Neurodegenerative Disorder
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurodegenerative disorders associated with sleep disorders
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Neuropsychological assessment, brain MRI, electroencephalogram and biomarker datas will be collected

SUMMARY:
Cognitive impairment often appears in neurodegenerative diseases, and it is expected to further study the mechanism of sleep disorders associated with the progression of neurodegenerative diseases by exploring the clinical manifestations, imaging, and biological marker changes of sleep disorders in neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of neurodegenerative disease.
2. patients experience insomnia, excessive drowsiness, or confusion at night.
3. Patients experience frequent awakenings, daily sleep episodes, or nocturnal confusion.
4. The presence of one or more of the following characteristics: a. wandering at night with inappropriate activity; b. agitation, combativeness; c. confusion, disorientation, or marked delirium.
5. Polysomnographic monitoring showed the following two conditions: a. poor sleep efficiency, increased number and duration of awakenings; b. multiple sleep latency tests showed increased daytime sleepiness.
6. Presence of other medical symptoms that do not indicate the primary disease.
7. Other sleep disorders (e.g., periodic limb movement disorders, obstructive sleep apnea syndrome) may be present, but do not explain the patient 's main symptoms.
8. any of the above can be diagnosed

Exclusion Criteria:

1. Patients with other neurological disorders.
2. Pregnant or lactating women.

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Neurodegenerative disorders are a cluster of chronic progressive diseases characterized by specific pathological manifestations. Common neurodegenerative disorders include Alzheimer's disease, Parkinson's disease and so on. We studied people with sleep disorders associated with neurodegenerative disorders.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
PSQI Scores | Baseline
  Pittsburgh Sleep Quality Index (PSQI),

SECONDARY OUTCOMES:
MoCA scores | Baseline
  The Montreal Cognitive Assessment (MoCA)
ACE-III scores | Baseline
  Addenbrooke's Cognitive Examination (ACE) score
HRV (ms) | Baseline
  Heart rate variability (HRV) was calculated as the maximum bpm - minimum bpm.
Plasma Aβ-42 levels (ng/ml) | Baseline
Vic | Baseline
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.
PAF (Hz) | Baseline
  The alpha-peak frequency (PAF) is the frequency with the highest power within the alpha-band.
Vic | 1 year after baseline
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No